CLINICAL TRIAL: NCT07250438
Title: Music Therapy Awareness in the Lecture Hall: Effects of Mindfulness-based Breathing and Core Exercises on Stress, Endurance, and Relaxation in University Students
Acronym: MT WİTH CORE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Emine Merve Ersever, Assistant Professor, Department of Physiotherapy and Rehabilitation, Ankara University, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-79176220-050.04-1961949; Ankara University (Other: ankara University)
Record Dates: First submitted 2025-09-30; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Stress in University Students; Relaxation and Well-being; Psychological Resilience
Keywords: Stress Management; Psychological Resilience; Mental Health and Well-being in University Students
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (No Intervention): Participants continue their usual activities without a structured program during the study period. Optionally, they may be offered the program after study completion
- Core exercise (Experimental): Participants in the experimental group receive a combined intervention including mindfulness-based breathing exercises, core stabilization training, and music therapy sessions for stress reduction and relaxation.
  Interventions: Behavioral: core exercise

INTERVENTIONS:
Behavioral: core exercise — Participants will engage in a structured program combining mindfulness-based breathing exercises, core stability/strength exercises, and music therapy awareness sessions. Sessions will be delivered in a lecture-hall setting, approximately 2-3 times per week, lasting 45-60 minutes, for a total duration of 4-8 weeks.
  Arms: Core exercise

SUMMARY:
This study aims to evaluate the effects of music therapy awareness, mindfulness-based breathing, and core exercises on stress, resilience, and relaxation in university students. Stress is highly prevalent in this population and can negatively affect both academic performance and physical and psychological health. By combining music therapy with breathing and core exercises, the study seeks to provide a holistic approach to improving students' well-being

DETAILED DESCRIPTION:
University students often experience high levels of stress due to academic and social responsibilities, which may lead to reduced cognitive performance, decreased endurance, and health problems. Effective stress management strategies are therefore essential to support academic achievement and quality of life.

Music therapy has been shown to reduce stress and promote relaxation. Mindfulness-based breathing exercises enhance body awareness, calmness, and resilience, while core exercises improve physical endurance, posture, and general well-being. In a university setting, the integration of these approaches may reduce stress levels and increase both psychological and physical resilience.

This study will recruit 80 healthy volunteers aged 18-30, consisting of university students or young adults. Participants must be willing to give informed consent and must not have severe musculoskeletal, neurological, or systemic health conditions that prevent exercise. Individuals with significant hearing loss, recent surgery, or psychiatric conditions that may interfere with participation will also be excluded.

The primary objective is to investigate the effects of music therapy awareness, mindfulness-based breathing, and core exercises on stress levels, resilience, and relaxation among students. The secondary objective is to explore the potential impact of these interventions on academic performance and social relationships.

ELIGIBILITY:
Inclusion Criteria:

* Healthy university students or young adults aged 18-30 years.
* Willing to participate voluntarily and able to provide written informed consent.
* major physical health problems or musculoskeletal injuries that would prevent participation in the exercise program, based on preliminary health screening.
* No significant hearing impairment that would interfere with participation in music-based sessions

Exclusion Criteria:

* Acute or chronic musculoskeletal pain, injury, or disorders that limit exercise participation.
* Serious cardiovascular, pulmonary, or other systemic diseases that restrict physical activity.
* History of surgery within the past 3 months or medical advice to avoid exercise
* Psychiatric or neurological disorders that may prevent compliance with the program.
* Significant hearing impairment or other sensory deficits that could interfere with music therapy sessions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived Stress Score assessed by the Perceived Stress Scale (PSS) | Baseline and 6 weeks
  The Perceived Stress Scale (PSS) is a 10-item self-report questionnaire designed to measure the degree to which individuals perceive their lives as stressful. Each item is rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often).
  Total scores range from 0 to 40, with higher scores indicating greater perceived stress
Change in core muscle endurance assessed by the Plank Test | Baseline and 6 weeks
  Core muscle endurance will be evaluated using the Plank Test. Participants are instructed to hold a standard prone plank position for as long as possible.
  The time (in seconds) is recorded from the start of the position until loss of proper form or voluntary termination.
Change in core muscle endurance assessed by the Plank Test assessing by score | Baseline and 6 weeks
  Core muscle endurance will be evaluated using the Plank Test. Scores range from 0 seconds (minimum) to the maximum duration the participant can maintain proper posture

SECONDARY OUTCOMES:
Change in relaxation/calmness assessed by 5-point Likert Scale questionnaire | Baseline and 6 weeks
  Participants rate their perceived relaxation on a 5-point Likert Scale (1 = very tense, 5 = very relaxed). Higher scores indicate greater calmness and relaxation (better outcome)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol